CLINICAL TRIAL: NCT05264350
Title: A Prospective, Multicenter, Randomized, Controlled, Blinded Post-Market Clinical Follow-up Investigation to Verify Clinical Efficacy, Performance, and Safety of Viiral® Nasal Spray, Compared to Control, When Used According to Intended Use in Subjects With Dry Nose Symptoms
Brief Title: A Post-Market Clinical Follow-up Investigation to Verify Performance and Safety of Viiral®Nasal Spray in Subjects With Dry Nose Symptoms
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Viiral Nordic AB (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Vii-001
Record Dates: First submitted 2022-02-03; First posted 2022-03-03 (Actual); Last update posted 2022-10-13 (Actual); Status verified 2022-10

CONDITIONS: Rhinitis Sicca

STUDY DESIGN:
Intervention Model Description: Subjects will be randomised in proportions 2:1, Viiral® Nasal Spray group: Isotonic Saline Nasal Spray group. Block randomisation will be performed with varying block sizes. Numbered randomisation envelopes containing cards with code numbers will be prepared.
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Viiral® Nasal Spray group (Experimental): The nasal spray to be administrated twice daily for 8 weeks.
  Interventions: Device: Sialic acid nasal spray
- Isotonic Saline Nasal Spray (Active Comparator): The nasal spray to be administrated twice daily for 8 weeks.
  Interventions: Device: Isotonic Saline Nasal Spray

INTERVENTIONS:
Device: Sialic acid nasal spray — The nasal spray will be self administered twice daily for 8 weeks.
  Arms: Viiral® Nasal Spray group
Device: Isotonic Saline Nasal Spray — The nasal spray will be self administered twice daily for 8 weeks.
  Arms: Isotonic Saline Nasal Spray

SUMMARY:
A chronic irritation of the nasal mucosa can be painful and unpleasant for the individual. Dry nasal mucosa with scabs is a common problem but not everyone seeks care. The causes can be several such as staying for long periods in dry and dusty air, hot rooms or hot environments, tobacco smoke, side effects of drugs and mechanical irritation (nasal congestion). The nasal spray contains salic acid (neuraminic acid). This substance is found naturally in humans in the nasal mucosa which keeps it moist. Salic acid is also found, for example, in breast milk and is also found in food production. Previous studies have shown that treatment with salic acid is gentle, relieves symptoms and has a soothing and moisturising effect.

The purpose of the study is to evaluate whether the symptoms of dry nose can be improved with treatment with Viiral®Nasal spray and have a soothing and moisturising effect. The treatment also aims to prevent colds caused by viruses.

As a control product in the study, a nasal spray with isotonic saline solution will be used. In this study, a total of 78 women and men who have been diagnosed with dry nose / rhinitis sicca will be included in the study. After the participants have given their consent to participate in the study, treatment with the study product or control product will begin. The treatment is started by the study participants themselves at home. Two thirds will be treated with the study product and one third will be treated with a control product. Clinic visits will be performed at three occasions after the screening/baseline visit, at day 14, day 28 and on day 56.

ELIGIBILITY:
Inclusion Criteria:

* Signed Informed Consent Form.
* Adult males and females ≥ 18 years old.
* Score of at least 10 as indication for application of moistening nasal sprays per investigator judgement, confirmed with a total Rhinitis Sicca Symptom Score (sensation of dry nose, nasal obstruction, crusting, itching/sneezing attacks, pain in the nose, runny nose, thick nasal discharge, dry throat, impairment of smell and impairment of sleep) using a 5-point severity scale (0=none, 1=mild, 2=moderate, 3=strong, and 4 = very strong.
* Able to use the device independently.

Exclusion Criteria:

* Antiallergy drugs and rhinitis medication, including rescue medication for symptom relief and anti-hyperactivity last week.
* Pregnancy or lactation at time of investigation participation.
* Physical or mental impairment affecting subjects' ability to use the device, per investigator judgement.
* Person not suitable for the investigation according to the investigator judgement.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2022-02-03 (Actual); Primary Completion 2022-08-16 (Actual); Study Completion 2022-09-15 (Actual)

PRIMARY OUTCOMES:
Rhinitis Sicca Symptom Score (RSSS) | Up to 8 weeks.
  RSSS score constitutes of the sum of ten (10) individual symptoms. Each symptom assessed on 5-point scale (0 = none, 1 = mild, 2 = moderated, 3 = strong, 4 = very strong).
  1. Sensation of dry nose
  2. Impairment of nasal breathing/nasal obstruction
  3. Crusting
  4. Itching/ sneezing attacks
  5. Pain in the nose
  6. Nasal discharge anterior/runny nose
  7. Thick nasal discharge
  8. Desire to clear one's throat /dry throat
  9. Impairment of smell
  10. Impairment of sleep

SECONDARY OUTCOMES:
Nasal spray sensory scale (NSSS) | Up to 8 weeks.
  Tolerability examination, sensory perception of the spray. Parameters to be answered using visual analog scale (VAS 0 = worst grading - 100 = best grading)
  1. Did product have any taste?
  2. Did product run out of nose? (amount)
  3. Did product run down throat? (amount)
  4. Did you feel discomfort when nozzle was inserted to your nose?
  5. Did product induce the urgency to sneeze?
Short Form 12 (SF-12) | Up to 8 weeks.
  SF-12 is a health-related quality of life questionnaire consisting of twelve questions that measure functional health and well-being form the subject's point of view.
Endoscopy score of the nasal cavity (ES) | Up to 8 weeks.
  Changes of the nasal mucosa using a 3-point scale (0 = no, 1 = mild, 2 = severe).
  1. Classification of crusting
  2. Dryness of mucosa
  3. Redness and oedema of nasal mucosa
  4. Atrophy
Episodes of common cold/sick days | Up to 8 weeks.
  The total number of common cold episodes and episodes days.

CONTACTS AND LOCATIONS:
Locations (2):
- Sweden (2):
  - Universitetssjukhuset, Avdelning för kliniska prövningar, Örebro, Region Örebro
  - Cordinator Medical Service AB, Linköping, Region Östergötland

IPD SHARING:
Plan to Share IPD: Undecided